CLINICAL TRIAL: NCT07097896
Title: Bronchoscopic Lung Volume Reduction With Endobronchial Silicone Valve for Patients With Emphysema: a Randomised Controlled Trial
Brief Title: Endobronchial Silicone Valve for Patients With Emphysema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Beijing Cardiotech Medical Technology CO., LTD (Unknown)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ESV-1
Record Dates: First submitted 2025-07-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Emphysema
Keywords: Endobronchial Lung Volume Reduction; Emphysema; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESV and Optimal Medical Management (Experimental): This study arm will undergo ESV treatment along with optimal medical management, including smoking cessation program, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Interventions: Device: ESV
- EBV and Optimal Medical Management (Other): This study arm will undergo EBV treatment along with optimal medical management, including smoking cessation program, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Interventions: Device: EBV

INTERVENTIONS:
Device: ESV — This study arm will undergo ESV treatment and also receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Arms: ESV and Optimal Medical Management
Device: EBV — This study arm will undergo EBV treatment and also receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Arms: EBV and Optimal Medical Management

SUMMARY:
The purpose of this research is to compare the efficacy and safety between endobronchial silicone valve and endobronchial valve in bronchoscopic lung volume reduction in patients with severe emphysema.

DETAILED DESCRIPTION:
The Cardiotech medical technology CO., LTD Endobronchial Silicone Valve (ESV) is a novel designed implantable bronchial valve intended to decrease volume in targeted regions of the lung. It is indicated for the treatment of patients with severe emphysema. The ESV are placed in the diseased region of the lung using bronchoscopy. Bronchoscopy is a way to access the lungs using a small tube with a camera on the end. As the diseased region of the lung shrinks in size, healthier regions may expand and function more efficiently, resulting in improved breathing.

This clinical trial included two groups. Participants are assigned at random to the 'Treatment' group or to the 'Control' group. The 'Treatment' group will receive the Cardiotech medical technology CO., LTD Endobronchial Silicone Valve (ESV) with optimal medical therapy. The 'Control' group will receive Zephyr Endobronchial Valve (EBV) in combination with optimal medical therapy. For every three participants in the study, two will go into the 'Treatment' group and one will go into the 'Control' group.

It is hypothesized that the ESV has similar efficacy and safety to EBV in treating patients with severe emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological evidence of emphysema
* Nonsmoking for 4 months prior to screening interview
* BMI less than 35 kg/m2
* Stable on current medication regimen
* Forced expiratory volume in one second (FEV1) between 15% and 45% of predicted value
* Residual Volume less than 175% predicted (determined by body plethysmography)
* Little or no collateral ventilation (CV-) as determined using the Chartis System

Exclusion Criteria:

* Had two or more hospitalizations over the last year for a COPD exacerbation
* Had two or more hospitalizations over the last year for pneumonia
* Had a prior lung transplant, lung volume reduction surgery, bullectomy or lobectomy
* Had a heart attack or congestive heart failure within the last 6 months
* Have heart arrhythmia
* Is alpha-1 antitrypsin deficient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1-second (FEV1) | 1-year
  Difference between study arms in absolute change from baseline for post-bronchodilator FEV1 score at 1 year (value at 1 year minus value at baseline).

SECONDARY OUTCOMES:
FEV1 Post-bronchodilator Absolute Change | 1 year
  Difference between study arms in absolute change from baseline for post-bronchodilator FEV1 score at 1 year (value at 1 year minus value at baseline).
St. George's Respiratory Questionnaire (SGRQ) | 1 year
  Difference between study arms in 'absolute change from baseline' for SGRQ score at 1 year (value at 1 year minus value at baseline).
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
6-minute Walk Distance | 1 year
  Difference between study arms in 'absolute and percentage change from baseline' for 6MWD at 1 year (value at 1 year minus value at baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No